CLINICAL TRIAL: NCT04293887
Title: Randomized, Open, Blank Control Study on the Efficacy and Safety of Recombinant Human Interferon α1β in the Treatment of Patients With New Type of Coronavirus Infection in Wuhan
Brief Title: Efficacy and Safety of IFN-α2β in the Treatment of Novel Coronavirus Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zhao Jianping, Director of Respiratory and Critical Care Medicine , Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zhaojp
Record Dates: First submitted 2020-02-15; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: COVID-19; Recombinant Human Interferon α1β
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard therapy + interferon therapy (Experimental): Standard treatment + recombinant human interferon α1β 10ug Bid was administered by nebulization for 10 days.
  Interventions: Drug: Recombinant human interferon α1β
- Standard therapy + blank therapy (No Intervention): Standard therapy

INTERVENTIONS:
Drug: Recombinant human interferon α1β — Saline needle 2ml + recombinant human interferon α1β10ug bid nebulization inhalation
  Arms: Standard therapy + interferon therapy

SUMMARY:
New coronavirus infection is an important cause of public health emergencies at home and abroad, which seriously affects people's health and social stability. The outbreak of SRAR-COV in China in 2003 caused serious social impact. From January 2002 to August 7, 2003, there were a total of 8,422 cases worldwide, involving 32 countries and regions, of which 919 cases were fatal, with a fatality rate of nearly 11%. The fatality rate of elderly patients and patients with underlying diseases was even more high.There is no precise and effective treatment for coronavirus infection. In vitro, IFN-α2β has inhibitory effects on MERS-CoV and closely related coronavirus severe acute respiratory syndrome (SARS) -CoV. A study showed the effects of interferon-α2β and ribavirin on the replication of nCoV isolates hCoV-EMC / 2012 in Vero and LLC-MK2 cells. The combined application may be useful for the management of patients with nCoV infection in the future. At present, the combination therapy of interferon α2β and ribavirin has been successfully applied in the initial treatment and prevention of SARS and MERS.The purpose of this study was to evaluate the efficacy and safety of recombinant human interferon α1β in treating patients with new coronavirus infection in Wuhan.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, open, blank-controlled, multi-stage clinical study. As there are no effective treatments, the project team will evaluate possible treatments (including but not limited to interferon α) based on actual conditions. , Lopinavir / ritonavir, remdesivir, single / polyclonal antibodies against coronavirus), explore the most effective antiviral treatment options.

The first phase will assess the efficacy and safety of interferon alpha compared to standard treatment for approximately 328 hospitalized adult patients diagnosed with a new coronavirus infection in Wuhan.

Patients with COVID-19 within 7 days of onset of symptoms were screened and randomly assigned as soon as possible after screening (within 24 hours). Patients will be allocated in a 1: 1 ratio, receiving the interferon alpha treatment group or only the standard treatment group. Patients who do not meet the inclusion and exclusion criteria are only allowed to be re-screened once, provided that the time from symptom onset to randomization remains within 7 days.

This study planned to randomize approximately 328 adult subjects. It will be stratified according to whether the onset time is ≤ 3 days, and randomly divided into groups of 1: 1, receiving standard treatment or interferon alpha atomization twice a day, 1 stick (10ug) each time, treatment course For 10 days. Subjects and all research center staff were not blinded.

The primary endpoint of this study was the incidence of side effects within 14 days of enrollment. Therefore, a 14-day visit is essential for the data needed for this endpoint. Every effort should be made to ensure that this study visit is completed in a timely manner.

Out-of-hospital treatment or discharge will reach the discharge standard on the day of implementation and will be implemented in accordance with the Health and Medical Commission's "Unknown Viral Pneumonia Diagnosis and Treatment Plan (Trial)". For patients treated outside the hospital or who have been discharged, final assessments are performed by phone and using a questionnaire (if applicable).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Clinically diagnosed patients with new type of coronavirus pneumonia, including: in accordance with the criteria for suspected cases, have one of the following etiology evidence:

   ① Real-time fluorescence RT-PCR of respiratory specimens or blood specimens for detection of new coronavirus nucleic acid;

   ② Sequencing of viral genes in respiratory specimens or blood specimens, highly homologous to known new coronavirus
3. The time interval between the onset of symptoms and random enrollment is within 7 days. The onset of symptoms is mainly based on fever. If there is no fever, cough, diarrhea or other related symptoms can be used.

Exclusion Criteria:

1. Any situation where the programme cannot be carried out safely;
2. Patients who have used interferon or remedesivir;
3. No clinical manifestations and chest imaging findings
4. Known allergy or hypersensitivity to interferon (including asthma);
5. Disabled in patients with uncontrolled autoimmune diseases;
6. Patients with severe heart disease, decompensated liver disease, renal insufficiency (CrCL <50ml / min), and those with abnormal bone marrow function are prohibited;
7. Epilepsy and impaired central nervous system function;
8. Pregnancy: Positive pregnancy test for women of childbearing age;
9. Breastfeeding women have not stopped breastfeeding;
10. The patient may be transferred to a non-participating hospital within 72 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of side effects | Within 14 days after enrollment
  dyspnea
The incidence of side effects | Within 14 days after enrollment
  SPO2≤94%
The incidence of side effects | Within 14 days after enrollment
  respiratory rate ≥24 breaths/min in oxygen state)

SECONDARY OUTCOMES:
Time from patient enrollment to clinical remission | Within 14 days after enrollment
  the patient had a normal body temperature of > for 24 hours (without taking antipyretic drugs or hormones) without self-consciousness Dyspnea or reduced dyspnea;
Proportion of patients with normal body | Within 14 days after enrollment
  Proportion of patients with normal body
Proportion of patients without dyspnea | Within 14 days after enrollment
  Proportion of patients without dyspnea
Proportion of patients without cough | Within 14 days after enrollment
  Proportion of patients without cough
Proportion | Within 14 days after enrollment
  Proportion of patients without oxygen treatment
The negative conversion rate of new coronavirus nucleic acid | Within 14 days after enrollment
  The negative conversion rate of new coronavirus nucleic acid
Proportion | within 28 days after enrollment
  Proportion of patients hospitalized/hospitalized in ICU
Frequency of serious adverse drug events. | within 28 days after enrollment
  Frequency of serious adverse drug events.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ksiazek TG, Erdman D, Goldsmith CS, Zaki SR, Peret T, Emery S, Tong S, Urbani C, Comer JA, Lim W, Rollin PE, Dowell SF, Ling AE, Humphrey CD, Shieh WJ, Guarner J, Paddock CD, Rota P, Fields B, DeRisi J, Yang JY, Cox N, Hughes JM, LeDuc JW, Bellini WJ, Anderson LJ; SARS Working Group. A novel coronavirus associated with severe acute respiratory syndrome. N Engl J Med. 2003 May 15;348(20):1953-66. doi: 10.1056/NEJMoa030781. Epub 2003 Apr 10. PMID 12690092
- [Background] Drosten C, Gunther S, Preiser W, van der Werf S, Brodt HR, Becker S, Rabenau H, Panning M, Kolesnikova L, Fouchier RA, Berger A, Burguiere AM, Cinatl J, Eickmann M, Escriou N, Grywna K, Kramme S, Manuguerra JC, Muller S, Rickerts V, Sturmer M, Vieth S, Klenk HD, Osterhaus AD, Schmitz H, Doerr HW. Identification of a novel coronavirus in patients with severe acute respiratory syndrome. N Engl J Med. 2003 May 15;348(20):1967-76. doi: 10.1056/NEJMoa030747. Epub 2003 Apr 10. PMID 12690091
- [Background] Fehr AR, Channappanavar R, Perlman S. Middle East Respiratory Syndrome: Emergence of a Pathogenic Human Coronavirus. Annu Rev Med. 2017 Jan 14;68:387-399. doi: 10.1146/annurev-med-051215-031152. Epub 2016 Aug 26. PMID 27576010
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Al-Tawfiq JA, Momattin H, Dib J, Memish ZA. Ribavirin and interferon therapy in patients infected with the Middle East respiratory syndrome coronavirus: an observational study. Int J Infect Dis. 2014 Mar;20:42-6. doi: 10.1016/j.ijid.2013.12.003. Epub 2014 Jan 6. PMID 24406736
- [Background] Falzarano D, de Wit E, Martellaro C, Callison J, Munster VJ, Feldmann H. Inhibition of novel beta coronavirus replication by a combination of interferon-alpha2b and ribavirin. Sci Rep. 2013;3:1686. doi: 10.1038/srep01686. PMID 23594967
- [Result] Falzarano D, de Wit E, Rasmussen AL, Feldmann F, Okumura A, Scott DP, Brining D, Bushmaker T, Martellaro C, Baseler L, Benecke AG, Katze MG, Munster VJ, Feldmann H. Treatment with interferon-alpha2b and ribavirin improves outcome in MERS-CoV-infected rhesus macaques. Nat Med. 2013 Oct;19(10):1313-7. doi: 10.1038/nm.3362. Epub 2013 Sep 8. PMID 24013700
- [Result] Kim UJ, Won EJ, Kee SJ, Jung SI, Jang HC. Combination therapy with lopinavir/ritonavir, ribavirin and interferon-alpha for Middle East respiratory syndrome. Antivir Ther. 2016;21(5):455-9. doi: 10.3851/IMP3002. Epub 2015 Oct 22. PMID 26492219
- [Result] Shalhoub S, Farahat F, Al-Jiffri A, Simhairi R, Shamma O, Siddiqi N, Mushtaq A. IFN-alpha2a or IFN-beta1a in combination with ribavirin to treat Middle East respiratory syndrome coronavirus pneumonia: a retrospective study. J Antimicrob Chemother. 2015 Jul;70(7):2129-32. doi: 10.1093/jac/dkv085. Epub 2015 Apr 21. PMID 25900158
- [Result] Min CK, Cheon S, Ha NY, Sohn KM, Kim Y, Aigerim A, Shin HM, Choi JY, Inn KS, Kim JH, Moon JY, Choi MS, Cho NH, Kim YS. Comparative and kinetic analysis of viral shedding and immunological responses in MERS patients representing a broad spectrum of disease severity. Sci Rep. 2016 May 5;6:25359. doi: 10.1038/srep25359. PMID 27146253